CLINICAL TRIAL: NCT03313011
Title: The Neurobiology of Two Distinct Types of Progressive Apraxia of Speech
Acronym: SLD4T
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Keith A. Josephs, Consultant in Neurology, Mayo Clinic
Other Study IDs: 17-002468
Record Dates: First submitted 2017-10-11; First posted 2017-10-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Apraxia of Speech; Non-fluent Aphasia; Primary Progressive Aphasia; Primary Progressive Nonfluent Aphasia
Keywords: apraxia of speech
MeSH Terms: conditions — Apraxias; Aphasia, Broca; Aphasia, Primary Progressive; Primary Progressive Nonfluent Aphasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will be asking for an optional blood sample to be stored and used for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Progressive Apraxia of Speech
  Interventions: Diagnostic Test: Testing protocol for the study

INTERVENTIONS:
Diagnostic Test: Testing protocol for the study — All patients will see a Neurologist for a neuro exam and consult, see a Speech Pathologist for assessment of speech and language skills, see the Study Coordinator for neuropsych testing (brief tests of thinking, memory, visual spatial skills, etc), undergo an MRI of the brain and a DaTscan of the brain.

SUMMARY:
The purpose of this study is to identify and distinguish two different types of Progressive Apraxia of Speech through clinical imaging and testing.

DETAILED DESCRIPTION:
Apraxia of speech (AOS) is a motor speech disorder reflecting a problem with the programming and/or planning of speech. AOS is well recognized in the context of stroke where onset is acute and the condition improves or is stable and chronic. AOS that is insidious in onset and progresses over time because of neurodegeneration is less well recognized and understood. For the past decade the investigators have been studying patients with primary progressive apraxia of speech (PAOS). They have demonstrated that it can be the earliest manifestation of an underlying neurodegenerative disease and have recently reported that the profile of PAOS characteristics can differ among affected patients. In some instances, the speech pattern is dominated by distorted sound substitutions and additions, and other features attributable to articulatory difficulty, while in other instances the pattern is dominated by slow, prosodically segmented speech. We have designated the first profile as Phonetic PAOS (Ph-PAOS) and the second as Prosodic PAOS (Pr-PAOS; previously referred to in our studies as type 1 and 2, respectively). Importantly, it appears that the AOS pattern type may have prognostic implications. In a recent longitudinal study, the investigators observed that in some PAOS patients, the AOS remained the most salient feature over an average of seven years of the neurodegenerative disease. Other patients developed a severe extrapyramidal syndrome, resembling progressive supranuclear palsy, within five years, causing significant morbidity, including the inability to ambulate and a shortened life span; interestingly, this more aggressive course was associated with the Pr- PAOS type. At present, little is known about these types. To address the main aim to better understand the neurobiology and clinical associations of PAOS types, they will perform longitudinal speech, language, and neurocognitive testing, acoustic analyses, neuroimaging, and autopsy in a cohort of 47 new PAOS patients (for 80 PAOS patients total) and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. All enrolled patients must be over the age of 18, speak English as their primary language, and have an informant who can provide an independent evaluation of functioning.
2. Each new patient must present with a chief complaint of progressive impairment of speech and must have evidence of AOS documented by a speech-language pathologist during routine clinical evaluation.
3. At study entry, all patients must have speech sufficiently intelligible for a confident diagnosis of AOS, dysarthria, and/or aphasia, and for acoustic analysis.

Exclusion Criteria:

1. Any patient whose speech is not intelligible enough for confident speech-language diagnosis will be excluded from the study.
2. All patients with concurrent illnesses that could account for speech deficits (e.g., traumatic brain injury, strokes, developmental syndromes), and patients meeting criteria for another neurodegenerative disease (e.g., Alzheimer's type dementia57), will be excluded.
3. Patients with aphasia or dysarthria who do not have PAOS, or whose aphasia or dysarthria at study entry is more severe than PAOS, will be excluded.
4. All women who are pregnant, or post-partum and breast-feeding, will be excluded as they are unable to undergo the required imaging. All women who can become pregnant must have a pregnancy test no more than 48 hours before the DaTscan.
5. Patients will also be excluded if MRI is contraindicated (e.g., metal in head, cardiac pace maker), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma or intracranial neoplasm), or if they are medically unstable or are on medications that might affect brain structure or metabolism (e.g. chemotherapy).
6. Patients will be excluded if they do not have an informant, or do not consent to the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have been diagnosed as having Progressive Apraxia of Speech.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Distinguish types of Progressive Apraxia of Speech | 1-2 years after baseline imaging
  Distinguish types of PAOS using the Apraxia of Speech Rating Scale (ASRS)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Josephs, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials